CLINICAL TRIAL: NCT03481387
Title: PERCEVAL S Valve Clinical Study for Chinese Registration
Acronym: PERFECT
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Corcym S.r.l (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TPS004
Record Dates: First submitted 2018-03-22; First posted 2018-03-29 (Actual); Last update posted 2024-03-06 (Actual); Status verified 2024-03

CONDITIONS: Aortic Valve Disease; Aortic Valve Stenosis
MeSH Terms: conditions — Aortic Valve Disease; Aortic Valve Stenosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Aortic Valve Replacement with Perceval S sutureless heart valve (Other): Patient undergoing Aortic Valve Replacement with Perceval S sutureless heart valve
  Interventions: Device: Aortic Valve Replacement with Perceval S sutureless heart valve

INTERVENTIONS:
Device: Aortic Valve Replacement with Perceval S sutureless heart valve — Patients will be treated with the PERCEVAL S heart valve (PERCEVAL S valve) which is a bioprosthesis manufactured with bovine pericardium and assembled on a Nitinol stent. The PERCEVAL S valve is designed to offer an alternative to surgically implanted flexible prostheses (stented and stentless biological valves). A special feature of the device is that it is self-anchoring and does not require sutures to be fixed to the implant site.

SUMMARY:
This is a prospective, open, single arm, multi-center clinical study in China. The primary objective of this study is to demonstrate the safety and effectiveness of the PERCEVAL S heart valve when used to replace a diseased native or malfunctioning prosthetic aortic valve in the indicated Chinese population for tissue heart valve replacement and suitable to the PERCEVAL S valve.

The secondary objectives are to collect all relevant device and subject demographics, procedural and hospital discharge, short and long-term data, as described in the secondary endpoints section.

ELIGIBILITY:
Inclusion Criteria:

1. Subject of age > 60 years.
2. Subject with aortic valve stenosis or steno-insufficiency.
3. Subject has signed the informed consent.
4. Subject in which preoperative evaluation is indicated for the need of native or prosthetic aortic valve replacement via open heart surgery
5. Subject is located in a geographic location that will enable the subject to return to the study site for follow-up examinations (i.e. geographically stable).

Exclusion Criteria:

1. Subject has preexisting valve prosthesis or annuloplasty rings in the mitral, pulmonic or tricuspid position.
2. Subject requires a double or multiple valve replacement or repair of the mitral, tricuspid, or pulmonic valve.
3. Subject requiring simultaneous cardiac procedures, apart from septal myectomy and/or coronary by-pass graft (CABG).
4. Subject has active endocarditis.
5. Subject has active myocarditis
6. Subject has aneurysmal dilation or dissection of the ascending aortic wall.
7. Subject is drug abuser, alcohol abuser, prison inmate, institutionalized, or is unable to give informed consent.
8. Subject has a major or progressive non-cardiac disease that, in the investigator's experience, results in a life expectancy of less than 1 year, or the implant of the device produces an unacceptable increased risk to the subject.
9. Subject with known hypersensitivity to nickel alloys.
10. Subject is undergoing renal dialysis for chronic renal failure or has hyperparathyroidism.
11. Subject has had an acute preoperative neurological deficit, myocardial infarction, or cardiac event that has not returned to baseline or stabilized for ≥30 days prior to the planned valve implant surgery.
12. Subject is known to be noncompliant or is unlikely to complete the study.
13. Subject with an aortic root enlargement, where the ratio between the diameter of the STJ and the annulus diameter, assessed by TEE, is > 1.3. Or for other anatomical reasons that not suitable for PERCEVAL S per IB.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2018-01-26 (Actual); Primary Completion 2020-09-25 (Actual); Study Completion 2024-02-25 (Estimated)

PRIMARY OUTCOMES:
composite endpoint of thromboembolism, all bleeding, all paravalvular leak and endocarditis, structural valve deterioration (SVD) and late all cause death (>30 days) | at one year
  The primary endpoint includes thromboembolism, all bleeding, all paravalvular leak and endocarditis, structural valve deterioration (SVD) and late all cause death (>30 days) per CEC adjudication
  The number and percentage of subjects with free from thromboembolism, all bleeding, all paravalvular leak and endocarditis, structural valve deterioration (SVD) and late all cause death will be presented, along with individual component of the success.

CONTACTS AND LOCATIONS:
Overall Officials: Sara Gaggianesi, Study Director — Corcym S.r.l
Locations (1):
- Fuwai Hospital CAMS&PUMC, Beijing, China

IPD SHARING:
Plan to Share IPD: Undecided